CLINICAL TRIAL: NCT03051945
Title: Endogenous Opioid Modulation by Ketamine
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Unable to perform brain imaging
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Brian Mickey, Principal Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 00087544
Record Dates: First submitted 2017-02-07; First posted 2017-02-14 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ketamine (Experimental): Ketamine will be infused via intravenous catheter over 40 minutes (0.75 mg/kg/hr over 40 minutes, 0.5 mg/kg total).
  Interventions: Drug: Ketamine Hydrochloride
- Placebo (Placebo Comparator): Normal saline will be infused via intravenous catheter over 40 minutes (0.75 mg/kg/hr over 40 minutes, 0.5 mg/kg total).
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Study drug will be infused while the participant sits or lies in a comfortable position. The dose of ketamine used does not cause unconsciousness but may cause perceptual disturbances.
  Arms: Ketamine
Other: Normal saline — Placebo
  Arms: Placebo

SUMMARY:
Demonstrate the acute effects of ketamine on endogenous µ-opioid neurotransmission in humans.

DETAILED DESCRIPTION:
This study will test the hypothesis that the rapidly-acting antidepressant ketamine improves core depressive symptoms by acutely activating the brain's endogenous µ-opioid system.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* DSM-5 major depressive disorder
* Current moderate-to-severe, treatment-resistant, depressive episode
* Patient Health Questionnaire (PHQ-9) total score ≥ 10
* PHQ-9 item score ≥ 2 on "Little interest or pleasure" item
* PHQ-9 item score ≥ 2 on "Feeling down, depressed, or hopeless" item
* Medical documentation of depression for at least 2 months
* Inadequate response to at least one adequate antidepressant medication trial in the current episode

Exclusion Criteria:

* Current episode duration >5 years
* Moderate-to-severe DSM-5 substance use disorder (past year)
* Cognitive disorder (past year)
* Post-traumatic stress disorder (past year)
* Obsessive compulsive disorder (past year)
* Personality disorder (past year)
* Positive urine drug screen
* Psychotic symptoms
* Mania
* Significant neurologic disorder or injury
* Breastfeeding or pregnancy
* Imminent suicide risk
* Current use of CYP3A4 inhibitors (e.g., ketoconazole or erythromycin)
* Other unstable psychiatric or medical condition requiring a higher level of care
* Contraindication to ketamine, MRI, or PET

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08 (Estimated); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale at 24 hours, change from baseline | 24 hr
  total score on the 17-item Hamilton Depression Rating Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No